CLINICAL TRIAL: NCT04105868
Title: Visuocortical Dynamics of Affect-Biased Attention in the Development of Adolescent Depression
Brief Title: Adolescent Attention to Emotion Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mary Woody, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY19010063; K23MH119225 (NIH)
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Results first posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurofeedback (Experimental): Participants will receive feedback about their attention to negative distractors during each trial using activity from their brain waves, which will help them reduce their attention to distractors.
  Interventions: Other: Neurofeedback

INTERVENTIONS:
Other: Neurofeedback — Participants will receive feedback during a computerized task that is based on their own visuocortical activity evoked by attention to negative distractors and task-relevant stimuli on the computer screen.

SUMMARY:
Rates of depression increase rapidly during adolescence, especially for girls, and, thus, research is needed to spur the development of novel interventions to prevent adolescent depression. This project seeks to determine if a novel visuocortical probe of affect-biased attention (i.e., steady-state visual evoked potentials derived from EEG) can 1) be used to prospectively predict depression using a multi-wave repeated measures design and 2) modify affect-biased attention and buffer subsequent mood reactivity using real time neurofeedback. This work could ultimately lead to improved identification of adolescents who are at high risk for depression and directly inform the development of mechanistic treatment targets to be used in personalized intervention prescriptions for high-risk youth.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include 90 female adolescents ages 13 years 0 months through 15 years 11 months at study entry.

Exclusion Criteria:

1. Lifetime history of any Diagnostic and Statistical Manual of Mental Disorders (DSM) 5 depressive disorder
2. Lifetime history of taking antidepressants [e.g., selective serotonin reuptake inhibitor (SSRIs)]
3. Lifetime history of a DSM 5 psychotic, bipolar, or autistic spectrum disorder.
4. Presence of EEG contraindications (e.g., personal lifetime history of seizures or family history of hereditary epilepsy).
5. Being pre-pubertal
6. Lifetime history of a neurological or serious medical condition.
7. Lifetime history of head injury or congenital neurological anomalies (based on parent report).
8. Intelligence quotient (IQ) less than 80, as assessed using the Wechsler Abbreviated Scale of Intelligence (WASI).
9. Uncorrected visual disturbance
10. Being acutely suicidal or at risk for harm to self or others.

Ages: 13 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2025-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Woody, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
We will comply with all National Institute of Mental Health (NIMH) guidelines regarding data repository/sharing.

REFERENCES:
- [Derived] Huang X, Mak J, Wears A, Price RB, Akcakaya M, Ostadabbas S, Woody ML. Using Neurofeedback from Steady-State Visual Evoked Potentials to Target Affect-Biased Attention in Augmented Reality. Annu Int Conf IEEE Eng Med Biol Soc. 2022 Jul;2022:2314-2318. doi: 10.1109/EMBC48229.2022.9871982. PMID 36085716

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Female adolescents aged 13-15 were recruited from the community to participate in a single-arm neurofeedback study on affect-biased attention. A total of 15 participants were enrolled.
Pre-assignment Details: All enrolled participants were assigned to the neurofeedback arm; no participants were excluded prior to assignment.
Period: Overall Study
Arm/Group | Neurofeedback
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All 15 participants assigned to the neurofeedback arm were included in the baseline analysis.
Arm/Group | Neurofeedback
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.67 (.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
SSVEP competition index [Mean (Standard Deviation); unit: Proportion (0-1)] — Competition indices for attention to the primary task vs. negative emotional distractors were calculated as the proportion of t-transformed SSVEP amplitudes to the task stimulus relative to the sum of amplitudes to both task and distractor stimuli (Task / [Task + Distractor]). Scores range from 0-1, with values above .50 reflecting greater attention to the task stimulus.
  Proportion (0-1) | .66 (.17)
Visual Analog Score - Sadness [Mean (Standard Deviation); unit: Score on 0-100 scale] — Participants rated their level of sadness on a Visual Analogue Scale (VAS) ranging from 0 = 'not at all' to 100 = 'extremely'. Scores reflect self-reported intensity of the emotional state at baseline. Population: One participant did not complete the baseline VAS Sadness measure, so data are reported for 14 participants.
  Score on 0-100 scale
    number analyzed (Participants) | 14
    (all) | 4.61 (12.72)
Visual Analog Score - Anxiety [Mean (Standard Deviation); unit: Score on 0-100 scale] — Participants rated their level of anxiety on a Visual Analogue Scale (VAS) ranging from 0 = 'not at all' to 100 = 'extremely'. Scores reflect self-reported intensity of the emotional state at baseline. Population: One participant did not complete the baseline VAS Anxiety measure, so data are reported for 14 participants.
  Score on 0-100 scale
    number analyzed (Participants) | 14
    (all) | 4.15 (6.59)

OUTCOME MEASURES:

1. Primary Outcome: Affect-biased Attention Following Neurofeedback (Immediately Post-Intervention)
Description: To measure affect-biased attention, steady-state visual evoked potentials (SSVEPs) were derived from EEG and used to index the amount of stimulus-driven attention to negative distractors relative to task-relevant stimuli. Affect-biased attention was assessed immediately before and immediately after the real-time SSVEP neurofeedback training to evaluate changes within the same session. The outcome below reflects the post-neurofeedback SSVEP competition index (Task / [Task + Distractor]). Scores above .50 indicate greater attention to the task stimulus.
Time Frame: Approximately 1 hour total: baseline assessment immediately before neurofeedback and post-neurofeedback assessment immediately after the ~1 hour training session on the same day.
Measure: Mean (Standard Deviation); unit: Proportion (0-1)
Arm/Group | Neurofeedback
Number analyzed (Participants) | 15
Proportion (0-1) | .41 (.18)
Statistical Analysis 1: Comparison: Neurofeedback; Null hypothesis: No within-subject change in SSVEP competition index from baseline to post-training; Test type: Other — Within-group pre/post differences were tested using a paired t-test; p = .004, t-test, 2 sided; Two-tailed paired samples t-test comparing baseline and post-training SSVEP competition index scores

2. Secondary Outcome: Sadness Ratings Following Laboratory Stressor (Immediately Post-Stressor)
Description: Participants completed a laboratory stressor following real-time SSVEP neurofeedback training to assess how well the intervention buffered sadness reactivity. State sadness was assessed immediately before and immediately after the stressor using a 100-millimeter visual analog scale (VAS) ranging from "neutral" to "very sad." Higher scores indicate greater sadness. The value reported below reflects the post-stressor rating.
Time Frame: Approximately 30 minutes total: baseline sadness rating immediately before and post-stressor rating immediately after the ~30-minute laboratory stressor on the same day.
Population: Three participants had missing VAS Sadness scores following the stressor.
Measure: Mean (Standard Deviation); unit: Score on 0-100 scale
Arm/Group | Neurofeedback
Number analyzed (Participants) | 12
Score on 0-100 scale | 2.80 (5.85)
Statistical Analysis 1: Comparison: Neurofeedback; Null hypothesis: No within-subject change in VAS Sadness scores from baseline to post-stressor; Test type: Other — Within-group pre/post differences were tested using a paired t-test; p = .25, t-test, 2 sided; Two-tailed paired samples t-test comparing baseline and post-stressor VAS sadness scores

3. Secondary Outcome: Anxiety Rating Following Laboratory Stressor (Immediately Post-Stressor)
Description: Participants completed a laboratory stressor following real-time SSVEP neurofeedback training to assess how well the intervention buffered sadness reactivity. State anxiety was assessed immediately before and immediately after the stressor using a 100-millimeter visual analog scale (VAS) ranging from "neutral" to "very anxious." Higher scores indicate greater anxiety. The value reported below reflects the post-stressor rating.
Time Frame: Baseline and following laboratory stressor (~30 minutes)
Population: Three participants had missing VAS anxiety ratings following the stressor.
Measure: Mean (Standard Deviation); unit: Score on 0-100 scale
Arm/Group | Neurofeedback
Number analyzed (Participants) | 12
Score on 0-100 scale | 3.29 (4.58)
Statistical Analysis 1: Comparison: Neurofeedback; Null hypothesis: No within-subject change in VAS Anxiety scores from baseline to post-stressor; Test type: Other — Within-group pre/post differences were tested using a paired t-test; p = .471, t-test, 2 sided; Two-tailed paired samples t-test comparing baseline and post-stressor VAS anxiety scores

ADVERSE EVENTS:
Time Frame: Single-session monitoring on the intervention day: from the start of baseline procedures (pre-neurofeedback) through 60 minutes after completion of the neurofeedback session; total monitoring duration ≈ 2 hours on the same day.
Description: Adverse events were monitored continuously during the above window via non-systematic assessment: spontaneous participant report and study-staff observation. Participants were queried at end-of-session and again at +60 minutes prior to discharge. No adverse events were observed or reported.
Arm/Group | Neurofeedback
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
The study was a small, single-arm pilot trial with 15 participants, which may limit generalizability. Results should be interpreted as preliminary pending replication in larger, controlled samples.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-23): https://cdn.clinicaltrials.gov/large-docs/68/NCT04105868/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT04105868/ICF_001.pdf